CLINICAL TRIAL: NCT01249313
Title: Risk Factor and Outcome of Candidemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chia Hui Chou, Division of Infectious Disease, China Medical University
Other Study IDs: DMR99-IRB-237
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Candidemia
Keywords: Risk; outcome
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Candidemia is the fourth leading cause of hospital-acquired infection in USA. In CMUH, it caused 9% hospital-acquired bloodstream infection in 2008 and 2009. In addition to increased mortality, candidemia also increased hospital stay and cost. There is a trend of increased cases of candidemia in recent years in CMUH. Early empirical and target treatment can reduce mortality and shortened length of hospital stay.

In the past, most prior studies in Taiwan dealt with risk factors for mortality rather than for candidemia and also focused at in vitro susceptibility to antifungal agents. In this study, the investigators hope to analyze the candidemic cases from 2003 to 2009, estimated 1000 cases. There were some rare Candida species. Therefore, the investigators hope to do case study for these diseases to provide the epidemiology of candidemia in CMUH. The result can help clinician in predicting the disease and its outcome. Besides, it also provides the epidemiology of candidemia in mid-Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* patient had candidemia from 2002-2010

Exclusion Criteria:

* no

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient had candidemia from 2002-2010
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-04 (Estimated); Study Completion 2012-12 (Estimated)